CLINICAL TRIAL: NCT05901922
Title: The Effect of Activity-Focused Social Skills Intervention on Praxis and Social Functioning in Individuals With Schizophrenia
Brief Title: The Effect of Social Skills Intervention on Praxis and Social Functioning in Individuals With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nigde Omer Halisdemir University (Other)
Responsible Party: Principal Investigator, Fatıma Zehra DOĞAN, lecturer, Nigde Omer Halisdemir University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NigdeOHU.OT
Record Dates: First submitted 2023-04-26; First posted 2023-06-13 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Schizophrenia
Keywords: schizophrenia; Social Skills; Apraxia, Motor; Social Functioning
MeSH Terms: conditions — Schizophrenia; Social Skills; Apraxias; Social Adjustment

STUDY DESIGN:
Intervention Model Description: 2 groups, an application and a control group, will be used. Social skills training will be applied to one of the two groups with schizophrenia and not to the other group.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Social skills training will be applied to this group. social skills training will be applied for 10 sessions. Sessions will be 2 sessions per week. Session duration will be 1 hour.
  Interventions: Behavioral: Social skills training
- control group (No Intervention): No intervention.

INTERVENTIONS:
Behavioral: Social skills training — In this training, role-playing will be done in groups of six. In these role playing, the importance and application of the social skill specified before the session will be studied.
  Arms: intervention group

SUMMARY:
This study will be carried out with individuals diagnosed with schizophrenia who continue to community mental health. Social skills training will be applied in the study. This study will be conducted to examine the effect of social skills training on praxis and social functionality in individuals with schizophrenia.

DETAILED DESCRIPTION:
This study will be conducted to examine the effect of social skills training on praxis and social functionality in individuals with schizophrenia. Test of Upper Limb Apraxia (TULIA) will be used for praxis assessment. Social Functioning Assessment Scale (SFAS) will be used for social functioning assessment. In this study, individuals with schizophrenia will be examined with the Model of Creativity Ability as an occupational therapy model and role playing activities will be determined according to the model. In secondary outcomes, the effect of social skills training on the symptoms of schizophrenia will be examined. therefore Scale for the Assessment of Positive Symptoms - SAPS and Scale for the Assessment of Negative Symptoms - SANS will be used in the study.

ELIGIBILITY:
Inclusion Criteria:

* Being an individual with a diagnosis of schizophrenia registered with the Community Mental Health Center
* Volunteering for the study and having written consent

Exclusion Criteria:

* Be under the age of 18 or over the age of 65
* Having a physical disability that limits participation in group activities

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-03-07 (Actual); Primary Completion 2023-06-10 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
The effect of social skills training on praxis in patients with schizophrenia was evaluated with TULIA | 2 months
  Test of Upper Limb Apraxia- TULIA: TULIA is a short-term apraxia test. TULIA was developed for the evaluation of hand movements (gestures) with and without symbolic meaning. Those that have symbolic value are also gestures associated with communication and also with the use of objects/tools. These three areas are evaluated as imitation (imitation) and pantomime ("pretending-following verbal instructions") examination by following the practitioner. Thus, TULIA, which consists of 6 subtests, consists of 48 items in the form of 8 items in each subtest. The 6-point scoring method (0-5) is used to calculate the result (range 0-240). A higher score means a better result in this assessment test. The test has Turkish validity.
The effect of social skills training on social functionality in individuals with schizophrenia | 2 months
  Social Functioning Evaluation Scale:This scale, which was developed in Turkey, evaluates social functioning in schizophrenia patients with 19 items and four sub-dimensions. Among the factors, interpersonal relations and entertainment consist of seven items, self-care consists of seven items, independent living skills consist of four items and work life consists of one item. The score that can be obtained from the scale is between 19 and 57, and a high score means a high level of social functionality.

SECONDARY OUTCOMES:
The effect of social skills training on schizophrenia positive symptoms in individuals with schizophrenia | 2 months
  Scale for the Assessment of Positive Symptoms - SAPS:
  The scale evaluates the level, distribution and severity of positive symptoms of patients with schizophrenia. The reliability of the Turkish form was made. It is a scale that has 4 subscales and includes 34 items. The subscales are hallucinations, delusions, strange behavior, and formal thought disorder. The scoring of each item varies between 0-5. The total score varies between 0-170. A lower score means a better result on this assessment test.
The effect of social skills training on schizophrenia negative symptoms in individuals with schizophrenia | 2 months
  Scale for the Assessment of Negative Symptoms - SANS:
  The scale evaluates the level, distribution and severity of negative symptoms of patients with schizophrenia. The reliability of the Turkish form was made. Has 5 subscales and includes 25 items. Subscales are affective blunting, alogy, apathy, anhedonia, and attention deficit. The scoring of each item varies from 0 to 25.The total score ranges from 0 to 125. A lower score means a better result on this assessment test.

CONTACTS AND LOCATIONS:
Overall Officials: Etem Erdal Erşan, professor, Study Director — Niğde Ömer Halisdemir University; Onur Altuntaş, associate professor, Study Director — Hacettepe University
Locations (1):
- Niğde Ömer Halisdemir University, Niğde, Bor, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No